CLINICAL TRIAL: NCT01775059
Title: Collection of Performance Data From the Integrated Sensor and Infusion Set. TRIAL 4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medtronic Diabetes R&D Denmark (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 277; 2012102304
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus Type I; Diabetes Mellitus Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

ARMS (1):
- Integrated sensor and infusion set. (Experimental)
  Interventions: Device: Integrated sensor and infusion set.

INTERVENTIONS:
Device: Integrated sensor and infusion set.

SUMMARY:
This is a multi-center, non-randomized, and interventional study in which subjects will use the Integrated sensor and infusion set with MiniLink Transmitter and the Medtronic Paradigm® VEO™ insulin pump (Sensor augmented pump) for 15 days.

The purpose of this study is to collect performance data on the Integrated sensor and infusion set for approximately 15 days, with the intention for each subject to wear 5 sets for 3 days each.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older at time of screening
* Subject has a clinical diagnosis of insulin requiring diabetes, as determined by investigator.
* Subject is currently using a Medtronic Paradigm Sensor Augmented insulin pump and has been so for a minimum of 3 months at time of enrollment.
* Subject has Continuous Glucose Monitoring experience (min 30% of CGM use within the month prior to enrollment).
* Subject has an average of 3 SMBG per day (verified via CareLink) during the month prior to enrollment.
* Subject is willing to wear the study devices for the duration of the study
* Subject is willing to perform frequent (min 7 per day) SMBGs during study device wear
* Subject is willing to keep a short diary during the device wear.

Exclusion Criteria:

* Female subject is pregnant, per urine pregnancy test performed at time of enrollment in women of child bearing age.
* Female subject plans to become pregnant during the course of the study.
* Subject is unable to tolerate tape adhesive in the area of the placement of the study device.
* Subject has any unresolved adverse skin condition in the area of the placement of the study device (e.g. psoriasis, rash, Staphylococcus infection).
* The subject is not deemed to be an appropriate candidate for the study by the investigator for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy endpoint | 5 months
  Agreement Rate (% within 20%) using VEO Pump
Safety endpoint | 5 months
  Descriptive summary of SAE, Adverse events and Device complaints

SECONDARY OUTCOMES:
Accuracy endpoint | 5 months
  Agreement Rate (% within 20%) using re-analyzed Guardian® REAL-Time and Paradigm® REAL-Time algorithm data

OTHER OUTCOMES:
Accuracy endpoint | 5 months
  MARD(%), BIAS(mg/dl), MAD(mg/dl) during study

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Pedersen-Bjergaard, MD, Principal Investigator — Hilleroed Hospital
Locations (3):
- Denmark (3):
  - Fredericia Hospital, Fredericia
  - Hilleroed Hospital, Hilleroed
  - Hvidovre Hospital, Hvidovre